CLINICAL TRIAL: NCT06099938
Title: Effect of Different Labour Analgesics on Maternal UtA, Fetal UA and MCA Blood Flow Index Observed by Doppler Ultrasonography：a Prospective Randomized Double-blinded Controlled Trial
Brief Title: Effect of Different Labour Analgesics on Maternal and Fetal Blood Flow Observed by Doppler Ultrasonography
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Yuqiong Liu, principal investigator, First Affiliated Hospital of Jinan University
Other Study IDs: june617
Record Dates: First submitted 2023-06-14; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Labor Pain; Analgesia; Fetus Disorder
Keywords: Sufentanil; Ropivacaine; Labor analgesia; Color Doppler ultrasound; Middle cerebral artery; Uterine artery; Umbilical artery
MeSH Terms: conditions — Labor Pain; Agnosia; Fetal Diseases | interventions — Sufentanil; Ropivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: intrathecal injections of sufentanil
  Interventions: Drug: sufentanil, ropivacaine
- Group R: intrathecal injections of ropivacaine
  Interventions: Drug: sufentanil, ropivacaine

INTERVENTIONS:
Drug: sufentanil, ropivacaine — The study used conventional anesthetic drugs to compare the effects of the two drugs on maternal and infant blood flow
  Other Names: Color Doppler ultrasound

SUMMARY:
Background: The purpose of this study was to see how intrathecal injections of sufentanil, ropivacaine, and sufentanil added to ropivacaine affected blood flow in the uterine artery, umbilical artery, and middle cerebral artery for combined spinal and epidural labor analgesia using color doppler ultrasound (CDUs).

Methods: A total of 90 singleton full-term parturients who were evaluated by obstetricians for feasible vaginal delivery were collected prospectively and divided into three groups based on the randomization and double-blind principle: sufentanil (S), ropivacaine (R) group, each with 30 cases. Main indicators include color doppler blood flow resistance indices (S/D) of the uterine artery (UtA), umbilical artery (UA), and middle cerebral artery (MCA) before (T0) and 30 minutes (T1), 60 minutes (T2), 90minutes (T3) after analgesia. Fetal heart rate (FHR), maternal mean arterial pressure (MAP) at T0, T1, T2 and T3。

DETAILED DESCRIPTION:
1. Randomization and blinding Parturients in the study were randomly assigned to Sufentanil group (S) and Ropivacaine group (R) by non-blind personnel according to the computer random number table, and the allocation was hidden. The solution was prepared by an unblinded anesthesiologist and packaged in a blind way and administered by another anesthesiologist. The patients, anesthesia providers, data recorders, ultrasound examiners, obstetrical staff, and nursing staff remained blinded to group assignment throughout the study.
2. Study intervention At the time of request for labor analgesia, patients were randomized to receive either sufentanil 5 μg (Group S) and ropivacaine 3mg (Group R) into the subarachnoid space. All groups received the standard epidural solution that contained 0.1% ropivacaine with 0.25 μg/ml sufentanil. Routine obstetric and anaesthetic monitoring was given after maternal entered the delivery room. An experienced the anesthesiologist select L3-4 lumbar vertebra clearance to puncture with standard sterile technique using loss of resistance when the puerpera palace has expanded to about 3 cm. After the puncture reached the epidural space, a 25-gauge lumbar anesthesia needle was used to puncture into the subarachnoid space. 2 mL of anesthetic drug as determined by her group randomization were administered into the cavity through the lumbar anesthesia needle after cerebrospinal fluid flow out. A 19-gauge spring-wound catheter was threaded 4-6 cm into the epidural space. All patients received a test dose of 3 ml of 1.5% lidocaine followed by an initial loading dose of 5 ml of the standard epidural solution. Epidural catheters into vessels or subarachnoid space were excluded. An analgesic pump (PCEA pump, 100ml) containing standard epidural solution was then connected to the epidural catheter at a background continuous infusion rate of 5 mL/h. The visual analogue score for pain (VAS) was performed 15 minutes after the injection dose, and if the VAS score fell below 3, the case was included in the study.

   An anesthesia provider assessed the adequacy of analgesia for the patients throughout the duration of labor. Any breakthrough pain was managed with a physician-administered epidural bolus. All obstetric analgesia procedures were performed by the same anesthesiologist to reduce errors due to technical reasons.
3. Ultrasonic examination method The patients were placed in a supine position with calm breathing to perform doppler ultrasonography during the interval of contractions. Ultrasound probe was placed on fetal head area. Middle cerebral arteries (MCA) run anteriorly on both sides of the ring of cerebral arteries at the position of the double head diameter (see Figure 1A). We can get waveforms of MCA examined by pulsed wave doppler (see Figure 1B). The probe was placed at the placenta area, and we can see the fetal umbilical cord connecting to the center of the placenta. Umbilical artery (UA) could be identified by color flow, and its waveforms were examined by pulsed wave doppler (see Figure 1C and 1D). The probe was placed at the midpoint of the groin. The right and left uterine arteries (UtA) could be identified by color flow at the apparent crossover with the external iliac arteries, and pulsed wave doppler was used to obtain waveforms (see Figure 1E and 1F). 3 to 10 arterial spectrograms with clear edges and no background noise at baseline were selected. The above arterial blood flow indexes were measured three times and the average value was taken. The S/Dvalue of MCA、UA、UtA can be measured automatically by ultrasound instrument. All doppler examinations were performed by the same sonographer.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade I to II
2. Aged 20 to 35 years
3. Weighing 50 to 100 kg
4. 150-175 cm in height
5. 37 to 41 weeks of gestation

Exclusion Criteria:

1. Women with contraindications of spinal anesthesia
2. Maternal complications (such as pregnancy-induced hypertension, preeclampsia, cardiovascular and cerebrovascular diseases, etc.)
3. Abnormal uterine contractions
4. Abnormal placental function or position
5. Signs of fetal distress
6. Known fetal malformations

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ASA grade I to II, aged 20 to 35 years, weighing 50 to 100 kg, 150-175 cm in height, and 37 to 41 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
color doppler blood flow resistance indices (S/D） | S/D measured before analgesia and 30 minutes, 60 minutes, 90minutes after analgesia
  S/D is an abbreviation for systolic/diastolic blood pressure.The patients were placed in a supine position with calm breathing to perform Doppler ultrasonography during the interval of contractions.

SECONDARY OUTCOMES:
FHR | Fetal heart rate measured before analgesia and 30 minutes, 60 minutes, 90minutes after analgesia
  Fetal heart rate
MAP | Mean arterial pressure before analgesia and 30 minutes, 60 minutes, 90minutes after analgesia
  Mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Xuemei Peng, Ph.d, Principal Investigator — First Affiliated Hospital of Jinan University
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT06099938/Prot_SAP_000.pdf